CLINICAL TRIAL: NCT01707875
Title: Fetal Brain Asymmetry: in Utero and Early Neonatal Follow up
Status: Terminated | Type: Observational
Why Stopped: Difficulties in recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: EMC-0062-12-CTIL
Record Dates: First submitted 2012-10-14; First posted 2012-10-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2012-07

CONDITIONS: Fetal Ventricle Brain Asymmetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fetal ventricle brain asymmetry
  Interventions: Other: fetal brain neurosonography

INTERVENTIONS:
Other: fetal brain neurosonography — fetal brain neurosonography according to the ISUG guidelines

SUMMARY:
Fetal brain asymmetry is considered a normal developmental processes. The size and shape of the lateral ventricles are interdependence with the brain parenchyma. Abnormal development of the fetal brain may cause unilateral or bilateral ventriculomegaly. Fetal cerebral ventricle measurement is one of the most frequently used sonographic tool for the evaluation of brain development. It is easier to evaluate and measure the distal cerebral ventricle, and therefore data concerning the normal range of asymmetry and the normal progress of the asymmetry are limited.

The objective of the study is to follow up the incidental finding of fetal ventricle brain asymmetry between 19-30 weeks of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 18-42 years old pregnant women
* 19-30 weeks of pregnancy
* No medical history of chronic disease
* No medical history of drug therapy
* No other findings on ultrasound examination
* Low risk pregnancy

Exclusion Criteria:

* Fetal malformation
* Chronic maternal disease
* Fetal chromosomal aberration
* suspected fetal infection

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with fetal ventricle brain asymmetry
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)